CLINICAL TRIAL: NCT03040505
Title: Future Mental Projections in Schizophrenia
Acronym: FutureProSchiz
Status: Terminated | Type: Observational
Why Stopped: The number of subjects needed was overestimated (from assumptions made in the litterature).
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6527
Record Dates: First submitted 2017-01-27; First posted 2017-02-02 (Estimated); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with schizophrenia: Patients with schizophrenia or schizoaffective disorder according to DSM-V criteria
  Interventions: Other: questionnary
- Control participants: - Control participants without psychiatric nor neurological history
  Interventions: Other: questionnary

INTERVENTIONS:
Other: questionnary — Participant's verbalization will be audio recorded and then transcribed by investigators. The investigators will use predefined categories to score the strategies mentioned by participants during the think aloud task.

SUMMARY:
The aim of the study is to investigate temporal organization of future thinking in patients with schizophrenia. Patients and control participants will be asked to envision and briefly describe ten personal future events using a cue-words list. Then they will be asked to describe everything that came to their minds (i.e. to think aloud) while they attempted to determine when an event will likely occur. The investigators will compare the proportion of several predefined strategies mentioned by the two groups of participants to locate future events in time. The investigators predict that patients will envision less personal future events and will rely to a lesser extent on strategies to locate events in time, than control participants.

ELIGIBILITY:
Inclusion Criteria:

* for patients only
* male or female
* age limits : 18-55 years old
* under the protection of health insurance
* who have signed up the consent form
* schizophrenia or schizo-affective disorder according to the DSM-5 criteria (APA, 2013).
* clinically stable for at least 2 months
* patients under guardianship or curatorship need agreement of their legal representative
* informed of the results of prior medical examination for controls only
* male or female
* age limits : 18-55 years old
* under the protection of health insurance
* who have sign up the consent form
* recruited from the general population and matched on gender, age years of schooling
* no psychiatric history (DSM-5)

Exclusion Criteria:

* for both patients and controls
* current severe or unstable somatic illness
* neurological history (brain injury > 15 minutes loss of consciousness , epilepsia, brain surgery…)
* current substance use disorder (DSM-5)
* current major depressive disorder (CDSS,BDI, HDRS)
* mental retardation (IQ < 70, WAIS-4, f-NART)
* history of general anesthesia 3 months prior to the experiment
* pregnancy declared by the subject
* breast feeding
* current legal control
* in emergency situation
* included during exclusion period in another experiment
* for controls only
* taking of antipsychotic drugs for the 3 weeks prior to inclusion
* under guardianship or curatorship

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients with Schizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2019-10-20 (Actual); Study Completion 2019-10-20 (Actual)

PRIMARY OUTCOMES:
Number of time location strategies | 1 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service de psychiatrie 1, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No